CLINICAL TRIAL: NCT01179282
Title: Repeated Nasal Challenge in Skin Prick-puncture Negative and Intradermal Positive Dust Mite Allergic Rhinitis Patients.
Acronym: DUSTMITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Richard Lockey, Principal Investigator, University of South Florida
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: intradermal positive dust mite
Record Dates: First submitted 2010-08-09; First posted 2010-08-11 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2013-01

CONDITIONS: ALLERGIC RHINITIS
Keywords: DUST MITE ALLERGIES
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PLACEBO (Placebo Comparator): PLACEBO NASAL SPRAY
  Interventions: Biological: dust mite extract or placebo
- DUST MITE ALLERGEN (Active Comparator): Subjects will use dust mite Dermatophagoides pteronyssinus (Dp) extract or placebo nasal spray at home for 2 weeks, with a 1 month washout period followed by 2 weeks of the other nasal spray.
  Interventions: Biological: dust mite extract or placebo

INTERVENTIONS:
Biological: dust mite extract or placebo — intervention will be to stop study drug or placebo

SUMMARY:
Subjects who have a clinical history of perennial rhinitis symptoms associated with dust exposure or not associated with other perennial allergens, will have a positive challenge with Dermatophagoides pteronyssinus. Subjects will be ppt negative and intradermal skin test positive to Dust p Challenges will be performed with placebo or Dp extract three times daily each for 2 weeks.

Primary endpoint after nasal challenge with Dust p Mean Symptom score increase by greater than or equal to 2 from baseline. Secondary Outcomes Mean decrease in PNIF by greater than 15percent from baseline. Mean increase in nasal lavage PGD2 and ECP by greater than 15percent from baseline levels.

Correlation between the orthogonol diameter of the wheal and flare of the intradermal skin test and the degree of symptom worsening during the nasal challenge.

These results will provide evidence for the continued use of the intradermal skin test in evaluating allergic rhinitis.

DETAILED DESCRIPTION:
All patients will be seen in the outpatient setting. After skin testing, subjects meeting established criteria will be placed in the study. Subjects will use dust mite Dermatophagoides pteronyssinus extract or placebo nasal spray at home for 2 weeks, with a 1 month washout period followed by 2 weeks of the other nasal spray. Both patients and investigators will be blinded as to which spray is being used. Subjects will monitor symptoms using a symptom score card and return to the research unit after the first and second week of challenge for review of symptoms and clinical assessment. If symptoms increase sufficiently to make the subject uncomfortable, they will return earlier. Testing will consist of peak nasal inspiratory flow rate and nasal lavage for PGD2 and ECP. Subjects will have these tests performed at the beginning of the study, and at the end of weeks 1 and 2.

One group of subjects will have a clinical history of perennial rhinitis symptoms associated with dust exposure or not associated with other perennial allergens. These subjects will be ppt negative and intradermal skin test positive to Dp. The other group of subjects will be the control group. They will be healthy with no history of rhinitis or rhinitis symptoms. They will be skin test negative. This group will also perform the same nasal challenge with placebo or Dp extract three times daily each for 2 weeks. This group will also perform the same tests as the rhinitis group.

In this study the research design is a prospective randomized double blind placebo controlled study. One addition is that both the experimental and control groups will use both types of nasal sprays, the Dp extract and the placebo during the nasal challenge. Each group will use one type of spray and then crossover to the other spray.

Study Population Inclusion Criteria Gender: Male or female Females are eligible to participate only if they are currently non-pregnant and non-lactating. Female subjects should not be enrolled if they plan to become pregnant during the time of the study.

Age: 18-65 years of age at enrollment Literacy: The subject must be able to read, comprehend, and record information in English.

Consent: The subject must have the ability to give informed consent. Type of subject: The subject must be seen in the outpatient setting. Skin test: The subject must be ppt negative and intradermal positive to Dp dust mite allergen defined by an orthogonal wheal 6 mm or greater than the saline negative control.

Rhinitis: The subject must have a history consistent with allergic rhinitis symptoms for at least 1 year.

Exclusion Criteria Ppt positive to major seasonal allergens; oak, cypress, cedar, Australian pine, or bayberry tree pollens.

Respiratory Instability: Hospitalization for respiratory disease within the last 6 months prior to entry into the study.

Respiratory Disease: Current diagnosis of asthma, cystic fibrosis, pneumonia, pneumothorax, atelectasis, pulmonary fibrotic disease, chronic bronchitis, or any other lower respiratory abnormalities.Respiratory Tract Infections: Confirmed or suspected infection of the nose, sinus, middle ear, oropharynx, upper respiratory tract, or lower respiratory tract within 28 days prior to testing.

Other Concurrent Conditions/Diseases: Any clinically significant, uncontrolled condition or disease state that, in the opinion of the investigator, would put the safety of the subject at risk through study participation or would confound the interpretation of the results if the condition/disease exacerbates during the study. The list of conditions/diseases that will result in exclusion if determined to be clinically significant includes, but is not limited to: cardiac arrhythmia; congestive heart failure; coronary artery disease; Addison's disease; diabetes mellitus; dyspnea; uncontrolled hypertension; hematological, hepatic, neurological, thyroid, peptic ulcer, or renal disease; immunologic compromise; current malignancy; or tuberculosis.

Physical Exam: Subjects who have nasal polyps, sinusitis, significant anatomic abnormality or infection of the upper airway will be excluded.

Recruitment Plan Screening will occur at participating clinical centers. Screening will include subjects listed in existing registries, referred by their healthcare professionals, and those who respond to IRB approved advertisements. Nasal symptom scores and demographic information will be verified, and the subject's interest in participating in the study will be discussed. Screening may take place in person or over the telephone.

Summary of visits for subjects Visit 1 Subjects will be given a symptom score card and calculate their baseline symptom score at home every night before bed for 7 days. (Table 2) Skin testing with DP dust mite allergen will be performed. Subjects who are ppt negative and intradermal positive will proceed. Subjects will complete a physical exam. (Table 1)

Visit 2 subjects with an average baseline symptom score less than 7 out of 15 total points will proceed.

Subjects will complete a physical exam. (Table 1) Baseline PNIF and nasal secretion collection will be performed in this order. Subjects will be assigned a nasal spray (placebo or dust) to be used at home three times daily in the morning, afternoon, and evening for 2 weeks and instructions will be given on its use.

Subjects will self-administer the nasal spray placebo or starting dose of Dp 500 AU/mL in each nostril under observation. If the challenge is positive by an increase in symptom score by greater than or equal to 3 from baseline; then PNIF and nasal secretion collection will be repeated after 15 minutes.

Subjects will be assigned a score card to record nasal symptoms before bed on each study day based on the previous 24 hours.

Visit 3 After 2 weeks of nasal spray usage subjects will return to the clinical research unit for testing consisting of PNIF and nasal secretion collection.

Subjects will return for testing any weekday during the 2 weeks if symptoms increase sufficiently to make them uncomfortable.

Nasal spray bottles will be weighed and symptom score card reviewed to monitor compliance.

Subjects will complete a physical exam. (Table 1) Visit 4 After 4 more weeks (the washout period); subjects will calculate their baseline symptom score at home every night before bed for 7 days.

On the 5th week subjects will return to the clinical research unit for a physical exam, baseline PNIF and nasal secretion collection.

Subjects will then be assigned (crossover) to the other nasal spray (placebo or Dp) to be used three times daily for 2 weeks with instructions given on its proper use.

Subjects will self-administer the nasal spray placebo or starting dose of D500 AU/mL in each nostril under observation. If the challenge is positive by an increase in symptom score by greater than or equal to 3 from baseline; then PNIF and nasal secretion collection will be repeated after 15 minutes.

Subjects will be assigned a score card to record nasal symptoms for the last 24 hours before bed on each study day Subjects will complete a physical exam. (Table 1) Visit 5 After 2 weeks of assigned nasal spray usage subjects will return to the clinical research unit for PNIF and nasal secretion collection.

Subjects will return for testing any weekday during the 2 weeks if symptoms increase sufficiently to make them uncomfortable.

Nasal spray bottles will be weighed and symptom score card reviewed to monitor compliance.

Subjects will complete a physical exam. (Table 1) Methods Skin Testing Medications known to affect skin test response will be withheld prior to testing. Ppt and intradermal testing will be done with Dp dust mite allergen, saline, and histamine controls. Criterion for a positive ppt result is a wheal diameter 3 mm or greater than the saline negative control. Criterion for a positive intradermal skin test result is a wheal 6 mm or greater than the saline negative control. Allergen and control skin tests are read at 15 minutes. Ppt will use standardized Dp (10,000 AU/mL; Greer Laboratories, Lenore, NC), glycerinated phenol saline (negative) and histamine (positive) controls (histamine base= 1.8 mg/mL) on the upper back. The minimum positive control will be a 3mm wheal diameter.

Intradermal testing on the upper arm will use standardized Dp (1,000 AU/mL; Greer Laboratories, Lenore, NC), glycerinated phenol saline (negative) and histamine (positive) controls (histamine base= 0.1 mg/mL; Greer Laboratories, Lenore, NC)

Testing technique Ppt: The GreerPick™ will be loaded with extract and inspected to ensure that a small droplet of extract is present at the tip of the device. While holding it at a 45 degree angle to the skin at the test site, the tip will be brought in contact with the skin. The tines will be pressed making contact with the superficial skin, withdrawing with a slight lifting of the skin. A properly applied prick test will result in a small pricking of the epidermis, but will not result in bleeding. The device will be discarded into a suitable biohazard container.

Intradermal testing: The volume of solution injected is 0.05mL. The disposable 0.5mL syringe with 27 gauge needle tip will be inserted at a 30 degree angle into the superficial skin layers. The solution will be injected maintaining steady pressure on the plunger until the volume is completely injected and the needle withdrawn. A distinct injection bleb should be observed. If leakage around the needle, an indistinct bleb or a subcutaneous injection occurs, then the test should be repeated at a different site. A tiny drop of extract at the injection site is common and will not affect test results.

Peak nasal inspiratory flow rate (PNIF) PNIF will be measured using the method described in the package insert for In-Check Nasal Inspiratory Flow Meter (Clement Clarke, Harlow, England Issue 2, 05/2000). The subject will exhale fully, hold the device horizontally, ensure the face mask forms an air tight seal around the nose, and inhale forcibly through the nose. This maneuver should be a short, sharp inspiratory action of about one-second duration. The test will be repeated 3 times and the highest result recorded. The clinical research unit staff will observe for possible obstruction called the nasal valve. This can occur during inspiration when the nostril(s) close and obstruct further inspiration. The test will be repeated if this occurs.

ELIGIBILITY:
Inclusion Criteria:

* Gender: Male or female
* Females are eligible to participate only if they are currently non-pregnant and non-lactating. Female subjects should not be enrolled if they plan to become pregnant during the time of the study.
* Age: 18-65 years of age at enrollment
* Literacy: The subject must be able to read, comprehend, and record information in English.
* Consent: The subject must have the ability to give informed consent.
* Type of subject: The subject must be seen in the outpatient setting.
* Skin test: The subject must be ppt negative and intradermal positive to Dp dust mite allergen defined by an orthogonal wheal 6 mm or greater than the saline negative control.
* Rhinitis: The subject must have a history consistent with allergic rhinitis symptoms for at least 1 year.

Exclusion Criteria:

* Ppt positive to major seasonal allergens; oak, cypress, cedar, Australian pine, or bayberry tree pollens.
* Respiratory Instability: Hospitalization for respiratory disease within the last 6 months prior to entry into the study.
* Respiratory Disease: Current diagnosis of asthma, cystic fibrosis, pneumonia, pneumothorax, atelectasis, pulmonary fibrotic disease, chronic bronchitis, or any other lower respiratory abnormalities.
* Respiratory Tract Infections: Confirmed or suspected infection of the nose, sinus, middle ear, oropharynx, upper respiratory tract, or lower respiratory tract within 28 days prior to testing.
* Other Concurrent Conditions/Diseases: Any clinically significant, uncontrolled condition or disease state that, in the opinion of the investigator, would put the safety of the subject at risk through study participation or would confound the interpretation of the results if the condition/disease exacerbates during the study. The list of conditions/diseases that will result in exclusion if determined to be clinically significant includes, but is not limited to: cardiac arrhythmia; congestive heart failure; coronary artery disease; Addison's disease; diabetes mellitus; dyspnea; uncontrolled hypertension; hematological, hepatic, neurological, thyroid, peptic ulcer, or renal disease; immunologic compromise; current malignancy; or tuberculosis.
* Physical Exam: Subjects who have nasal polyps, sinusitis, significant anatomic abnormality or infection of the upper airway will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2009-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Mean Symptom score increase by greater than or equal to 2 from baseline | at last study visit

SECONDARY OUTCOMES:
Mean increase in nasal lavage PGD2 and ECP by greater than 15 percent | last study visit
  Mean increase in nasal lavage PGD2 and ECP by greater than 15 percent from baseline levels. Correlation between the orthogonol diameter of the wheal and flare of the intradermal skin test and the degree of symptom worse

CONTACTS AND LOCATIONS:
Locations (1):
- Usf Asthma Allergy and Immunology Cru, Tampa, Florida, United States